CLINICAL TRIAL: NCT06413277
Title: Targeting the Conus Medullaris With ECAP-Controlled Closed-Loop SCS for the Treatment of Chronic Pelvic Pain: HOPE Trial
Brief Title: Targeting the Conus Medullaris With ECAP-Controlled Closed-Loop SCS for Treatment of Chronic Pelvic Pain: HOPE Trial
Status: Recruiting | Type: Observational
Sponsor: Ainsworth Institute of Pain Management (Other)
Collaborators: Saluda Medical Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 1351927
Record Dates: First submitted 2024-04-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pelvic Pain; Pudendal Neuralgia
Keywords: Chronic Pelvic Pain; Pudendal Neuralgia; Levator Ani Syndrome
MeSH Terms: conditions — Pudendal Neuralgia; Levator syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Saluda Evoke Smart SCS System — Surgical implantation of the Saluda Evoke Smart SCS System targeting the conus medullaris for stimulation

SUMMARY:
The aim of the study is to evaluate the effectiveness of using ECAP (electrically evoked compound action potential)-controlled CL (closed-loop) SCS (spinal cord stimulation) to treat chronic pelvic pain by stimulating an area in the spine called the conus medullaris (the lowermost tapering extremity of the spinal cord).

DETAILED DESCRIPTION:
Primary Objective Evaluate the efficacy of ECAP CL-SCS in treating chronic pelvic pain.

Secondary Objectives Evaluate changes in impact of pain on activities of daily living, pain quality, quality of life, sleep, anxiety and depression, pain catastrophizing, patient satisfaction, and symptoms related to urinary urgency frequency.

Evaluate safety of using ECAP-controlled CL-SCS in treating chronic pelvic pain. Summarize and evaluate device performance and typical programming parameters.

Study design This protocol describes an observational, prospective, single-arm, single center study. Eligible subjects will undergo an implant procedure as per standard of care for SCS. The system will be used within its licensed use. Data will be collected prospectively from 1 US study center. Time points of data collection are at baseline, trial, device implant and at 3-, 6-, -12 months post-implant.

Study population Subjects with chronic, intractable pelvic pain will be screened for participation in this study.

Subjects who provide informed consent and meet the study eligibility criteria will be enrolled and will undergo a trial procedure.

Following the trial phase subjects may receive a permanent implant and be followed up at 3-, 6-, and 12-months following the permanent implant.

Enrollment will continue until 15 subjects receive a permanent implant. We estimate that up to 20 subjects will be enrolled in this study.

Statistical analyses will be conducted using an appropriate software package (e.g., SAS, SPSS, R, Statistics). Standard summary statistics will be used to summarize endpoints and key study variables. Categorical variables, including the incidence of adverse events, will be summarized via counts and percentages. Continuous variables will be summarized via mean, median, standard deviation, and range. 95% confidence intervals will also be included with summary statistics for primary and secondary endpoints as well as other variables where appropriate. Any p-values for secondary or other endpoints will be nominal and not adjusted for multiplicity.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years of age or older at the time of enrollment.
2. Subject has a minimum Visual Analog Scale (VAS) score of 60 mm or higher (where 100 mm pain) at baseline.
3. Subject has been diagnosed with chronic intractable pain of the trunk and/or limbs specifically related to pelvic/genital/perineal/anorectal pain, which has been refractory to conservative therapy for a minimum of 6 months.
4. Subject has pain resulting from a known injury (surgery or trauma).
5. Subject has been clinically diagnosed with chronic pelvic pain (pain that occurs in the region of the pelvis), including diagnoses such as, but not limited to, complex regional pain syndrome (CRPS types 1 and 2), postsurgical pain, post-traumatic injury pain, interstitial cystitis/painful bladder syndrome, post-hysterectomy pain, post-prostatectomy pain, vulvodynia, chronic ovarian pain, and pudendal neuralgia of a known cause.
6. Subject is an appropriate candidate for the surgical procedures required in this study based on the clinical judgment of the implanting physician.
7. Subject is willing and capable of giving informed consent.
8. Subject is willing and able to comply with study-related requirements, procedures, and visits.

Exclusion Criteria:

1. Subject is pregnant or nursing.
2. Subject is involved in a malignancy or injury claim under current litigation or has pending/approved worker's compensation claim.
3. Subject's mechanism of pain is unknown.
4. Suspected cause and onset of pain are more than 30 days apart.
5. Subject has history of small fiber neuropathy, mitochondrial disease, fibromyalgia, addiction, CRPS in secondary pain area, and/or atypical facial pain.
6. Subject has been diagnosed with Crohn's Disease, Irritable Bowel Syndrome, ulcerous colitis, or any other inflammatory disease that is ongoing.
7. Subject has a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, as determined by the Investigator.
8. Subject has a history of sexual abuse and/or sexual trauma.
9. Subject has a history of unmanaged depression or anxiety that pre-dates the onset of symptoms.
10. Subject is using greater than 100 MME (morphine milligram equivalents) of opioids at baseline.
11. Subject shows evidence of an active, disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance of intervention, and/or ability to evaluate treatment outcomes.
12. Subject has previous neuromodulation experience including SCS (Spinal Cord Stimulator) and/or DRG (Dorsal Root Ganglion).
13. Subject has an existing drug pump and/or SCS system, or another active implantable device such as a pacemaker, deep brain stimulator, or sacral nerve stimulator.
14. Subject is concomitantly participating in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 or older with chronic, intractable pelvic pain
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Proportion of patients achieving at least 50% and 80% relief from pelvic pain and pelvic pain-related negative impact to quality of life compared to baseline | 12 months
  Pelvic Pain Reduction will be evaluated using the Visual Analog Scale (VAS) by comparing baseline VAS Scores to 3-, 6-, and 12- month post ECAP CL-SCS Implant VAS Scores.

SECONDARY OUTCOMES:
Impact of pain on activities of daily living: Proportion of patients achieving at least 50% and 80% reduction in impact of pain on activities of daily living compared to baseline. | 12 months
  Evaluate changes in impact of pain on activities of daily living from baseline to 3-, 6-, and 12-month post ECAP CL-SCS Implant using Pain Disability Index (PDI).
Changes in Pain quality: Proportion of patients achieving at least 50% and 80% relief in regard to pain quality compared to baseline | 12 months
  Evaluate changes in Pain quality from baseline to 3-, 6-, and 12-month post ECAP CL-SCS Implant using the Short Form-McGill Pain Questionnaire-2 (SF-MPQ2).
Changes in Health-Related Quality of life: Proportion of patients achieving at least 50% and 80% improvement in health-related quality of life compared to baseline. | 12 months
  Evaluate changes in health-related quality of life from baseline to 3-, 6-, and 12-month post ECAP CL-SCS Implant using EQ-5D-5L (The EuroQol 5 Dimension 5 Level self-report survey).
Changes in sleep quality: Proportion of patients achieving at least 50% and 80% improvement in sleep quality compared to baseline. | 12 months
  Evaluate changes in sleep quality and disturbances from baseline to 3-, 6-, and 12-month post ECAP CL-SCS Implant using Pittsburgh Sleep Quality Index (PSQI) questionnaire.
Changes in Anxiety and Depression: Proportion of patients achieving at least 50% and 80% reduction in anxiety and depression compared to baseline. | 12 months
  Evaluate changes in Anxiety and Depression from baseline to 3-, 6-, and 12-month post ECAP CL-SCS Implant using Hospital Anxiety and Depression Scale (HADS).
Changes in Pain Catastrophizing: Proportion of patients achieving at least 50% and 80% reduction in pain catastrophizing compared to baseline. | 12 months
  Evaluate changes in Pain Catastrophizing from baseline to at 3-, 6-, and 12-month post ECAP CL-SCS Implant using Pain Catastrophizing Scale (PCS).
Global Improvement: Proportion of patients achieving at least 50% and 80% increase in global improvement compared to baseline. | 12 months
  Evaluate changes in Global improvement with treatment at 3-, 6-, and 12-month post ECAP CL-SCS Implant using Patient global impression of change (PGIC) questionnaire.
Changes in Urinary Urgency Frequency: Proportion of patients achieving at least 50% and 80% reduction of urinary urgency frequency compared to baseline. | 12 months
  Evaluate changes in Urinary Urgency Frequency Patient Symptoms from baseline to 3-, 6-, and 12- month post ECAP CL-SCS Implant using Pelvic Pain and Urinary Urgency Frequency (PUF) Patient Symptom Scale.
Safety of ECAP CL-SCS: Number of participants who experience study-related adverse events (AEs) and serious AEs (SAEs), the seriousness and severity of the AEs/SAEs and how the AEs/SAEs relate to procedure, device, and/or stimulation. | 12 months
  Evaluate safety of ECAP CL-SCS in treating chronic pelvic pain by analyzing the incidence of study-related adverse event (AE) and serious AE (SAE).
Optimal device settings: Device settings at which participants achieved at least 50% and 80% increase in global improvement compared to baseline. | 12 months
  Device settings and data (e.g., ECAP target, amplitude, pulse width, frequency, programmed electrodes, recharge characteristics and patient usage) will be collected and summarized at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Corey W Hunter, MD, FIPP, Principal Investigator — Ainsworth Institute of Pain Management
Locations (1):
- Ainsworth Institute of Pain Management, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunter CW, Falowski S. Neuromodulation in Treating Pelvic Pain. Curr Pain Headache Rep. 2021 Feb 3;25(2):9. doi: 10.1007/s11916-020-00927-y. PMID 33534006
- [Background] Hunter CW, Stovall B, Chen G, Carlson J, Levy R. Anatomy, Pathophysiology and Interventional Therapies for Chronic Pelvic Pain: A Review. Pain Physician. 2018 Mar;21(2):147-167. PMID 29565946
- [Background] Gaskin DJ, Richard P. The economic costs of pain in the United States. J Pain. 2012 Aug;13(8):715-24. doi: 10.1016/j.jpain.2012.03.009. Epub 2012 May 16. PMID 22607834
- [Background] Fayaz A, Croft P, Langford RM, Donaldson LJ, Jones GT. Prevalence of chronic pain in the UK: a systematic review and meta-analysis of population studies. BMJ Open. 2016 Jun 20;6(6):e010364. doi: 10.1136/bmjopen-2015-010364. PMID 27324708
- [Background] Schappert SM, Burt CW. Ambulatory care visits to physician offices, hospital outpatient departments, and emergency departments: United States, 2001-02. Vital Health Stat 13. 2006 Feb;(159):1-66. PMID 16471269
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Korwisi B, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. Chronic pain as a symptom or a disease: the IASP Classification of Chronic Pain for the International Classification of Diseases (ICD-11). Pain. 2019 Jan;160(1):19-27. doi: 10.1097/j.pain.0000000000001384. PMID 30586067
- [Background] Stein SL. Chronic pelvic pain. Gastroenterol Clin North Am. 2013 Dec;42(4):785-800. doi: 10.1016/j.gtc.2013.08.005. Epub 2013 Oct 23. PMID 24280400
- [Background] Smith CP. Male chronic pelvic pain: An update. Indian J Urol. 2016 Jan-Mar;32(1):34-9. doi: 10.4103/0970-1591.173105. PMID 26941492
- [Background] Valovska, A. T. Pelvic Pain Management. (Oxford University Press, 2016).
- [Background] Mathias SD, Kuppermann M, Liberman RF, Lipschutz RC, Steege JF. Chronic pelvic pain: prevalence, health-related quality of life, and economic correlates. Obstet Gynecol. 1996 Mar;87(3):321-7. doi: 10.1016/0029-7844(95)00458-0. PMID 8598948
- [Background] Engeler DS, Baranowski AP, Dinis-Oliveira P, Elneil S, Hughes J, Messelink EJ, van Ophoven A, Williams AC; European Association of Urology. The 2013 EAU guidelines on chronic pelvic pain: is management of chronic pelvic pain a habit, a philosophy, or a science? 10 years of development. Eur Urol. 2013 Sep;64(3):431-9. doi: 10.1016/j.eururo.2013.04.035. Epub 2013 Apr 28. PMID 23684447
- [Background] Miller-Matero LR, Saulino C, Clark S, Bugenski M, Eshelman A, Eisenstein D. When treating the pain is not enough: a multidisciplinary approach for chronic pelvic pain. Arch Womens Ment Health. 2016 Apr;19(2):349-54. doi: 10.1007/s00737-015-0537-9. Epub 2015 May 5. PMID 25941014
- [Background] Lorencatto C, Petta CA, Navarro MJ, Bahamondes L, Matos A. Depression in women with endometriosis with and without chronic pelvic pain. Acta Obstet Gynecol Scand. 2006;85(1):88-92. doi: 10.1080/00016340500456118. PMID 16521687
- [Background] Williams DA. The importance of psychological assessment in chronic pain. Curr Opin Urol. 2013 Nov;23(6):554-9. doi: 10.1097/MOU.0b013e3283652af1. PMID 24080806
- [Background] Romao AP, Gorayeb R, Romao GS, Poli-Neto OB, dos Reis FJ, Rosa-e-Silva JC, Nogueira AA. High levels of anxiety and depression have a negative effect on quality of life of women with chronic pelvic pain. Int J Clin Pract. 2009 May;63(5):707-11. doi: 10.1111/j.1742-1241.2009.02034.x. PMID 19392920
- [Background] Yosef A, Allaire C, Williams C, Ahmed AG, Al-Hussaini T, Abdellah MS, Wong F, Lisonkova S, Yong PJ. Multifactorial contributors to the severity of chronic pelvic pain in women. Am J Obstet Gynecol. 2016 Dec;215(6):760.e1-760.e14. doi: 10.1016/j.ajog.2016.07.023. Epub 2016 Jul 18. PMID 27443813
- [Background] Martin CE, Johnson E, Wechter ME, Leserman J, Zolnoun DA. Catastrophizing: a predictor of persistent pain among women with endometriosis at 1 year. Hum Reprod. 2011 Nov;26(11):3078-84. doi: 10.1093/humrep/der292. Epub 2011 Sep 7. PMID 21900393
- [Background] McPeak AE, Allaire C, Williams C, Albert A, Lisonkova S, Yong PJ. Pain Catastrophizing and Pain Health-Related Quality-of-Life in Endometriosis. Clin J Pain. 2018 Apr;34(4):349-356. doi: 10.1097/AJP.0000000000000539. PMID 28731958
- [Background] Allaire C, Williams C, Bodmer-Roy S, Zhu S, Arion K, Ambacher K, Wu J, Yosef A, Wong F, Noga H, Britnell S, Yager H, Bedaiwy MA, Albert AY, Lisonkova S, Yong PJ. Chronic pelvic pain in an interdisciplinary setting: 1-year prospective cohort. Am J Obstet Gynecol. 2018 Jan;218(1):114.e1-114.e12. doi: 10.1016/j.ajog.2017.10.002. Epub 2017 Oct 12. PMID 29031895
- [Background] Carey ET, Martin CE, Siedhoff MT, Bair ED, As-Sanie S. Biopsychosocial correlates of persistent postsurgical pain in women with endometriosis. Int J Gynaecol Obstet. 2014 Feb;124(2):169-73. doi: 10.1016/j.ijgo.2013.07.033. Epub 2013 Oct 31. PMID 24290537
- [Background] Hunter C, Dave N, Diwan S, Deer T. Neuromodulation of pelvic visceral pain: review of the literature and case series of potential novel targets for treatment. Pain Pract. 2013 Jan;13(1):3-17. doi: 10.1111/j.1533-2500.2012.00558.x. Epub 2012 Apr 23. PMID 22521096
- [Background] Janicki TI. Chronic pelvic pain as a form of complex regional pain syndrome. Clin Obstet Gynecol. 2003 Dec;46(4):797-803. doi: 10.1097/00003081-200312000-00009. No abstract available. PMID 14595221
- [Background] Baranowski AP. Chronic pelvic pain. Best Pract Res Clin Gastroenterol. 2009;23(4):593-610. doi: 10.1016/j.bpg.2009.04.013. PMID 19647692
- [Background] Ploteau S, Labat JJ, Riant T, Levesque A, Robert R, Nizard J. New concepts on functional chronic pelvic and perineal pain: pathophysiology and multidisciplinary management. Discov Med. 2015 Mar;19(104):185-92. PMID 25828522
- [Background] Lee RB, Stone K, Magelssen D, Belts RP, Benson WL. Presacral neurectomy for chronic pelvic pain. Obstet Gynecol. 1986 Oct;68(4):517-21. PMID 3748502
- [Background] Ingber MS, Peters KM, Killinger KA, Carrico DJ, Ibrahim IA, Diokno AC. Dilemmas in diagnosing pelvic pain: multiple pelvic surgeries common in women with interstitial cystitis. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Mar;19(3):341-5. doi: 10.1007/s00192-007-0453-2. Epub 2007 Sep 18. PMID 17876490
- [Background] Udoji MA, Ness TJ. New directions in the treatment of pelvic pain. Pain Manag. 2013 Sep;3(5):387-94. doi: 10.2217/pmt.13.40. PMID 24654872
- [Background] Buffenoir K, Rioult B, Hamel O, Labat JJ, Riant T, Robert R. Spinal cord stimulation of the conus medullaris for refractory pudendal neuralgia: a prospective study of 27 consecutive cases. Neurourol Urodyn. 2015 Feb;34(2):177-82. doi: 10.1002/nau.22525. Epub 2013 Nov 19. PMID 24249588
- [Background] Fritz J, Chhabra A, Wang KC, Carrino JA. Magnetic resonance neurography-guided nerve blocks for the diagnosis and treatment of chronic pelvic pain syndrome. Neuroimaging Clin N Am. 2014 Feb;24(1):211-34. doi: 10.1016/j.nic.2013.03.028. Epub 2013 Aug 1. PMID 24210321
- [Background] Hayek SM, Veizi E, Hanes M. Treatment-Limiting Complications of Percutaneous Spinal Cord Stimulator Implants: A Review of Eight Years of Experience From an Academic Center Database. Neuromodulation. 2015 Oct;18(7):603-8; discussion 608-9. doi: 10.1111/ner.12312. Epub 2015 Jun 5. PMID 26053499
- [Background] Levine AB, Parrent AG, MacDougall KW. Stimulation of the Spinal Cord and Dorsal Nerve Roots for Chronic Groin, Pelvic, and Abdominal Pain. Pain Physician. 2016 Jul;19(6):405-12. PMID 27454271
- [Background] Saifuddin A, Burnett SJ, White J. The variation of position of the conus medullaris in an adult population. A magnetic resonance imaging study. Spine (Phila Pa 1976). 1998 Jul 1;23(13):1452-6. doi: 10.1097/00007632-199807010-00005. PMID 9670396
- [Background] Nashold BS Jr, Grimes J, Friedman H, Semans J, Avery R. Electrical stimulation of the conus medullaris in the paraplegic. A 5-year review. Appl Neurophysiol. 1977-1978;40(2-4):192-207. doi: 10.1159/000102443. PMID 309311
- [Background] Kapural L, Narouze SN, Janicki TI, Mekhail N. Spinal cord stimulation is an effective treatment for the chronic intractable visceral pelvic pain. Pain Med. 2006 Sep-Oct;7(5):440-3. doi: 10.1111/j.1526-4637.2006.00165.x. PMID 17014604
- [Background] Simopoulos T, Yong RJ, Gill JS. Treatment of Chronic Refractory Neuropathic Pelvic Pain with High-Frequency 10-kilohertz Spinal Cord Stimulation. Pain Pract. 2018 Jul;18(6):805-809. doi: 10.1111/papr.12656. Epub 2018 Jan 11. PMID 29106051
- [Background] Gorecki JP, Burt T, Wee A. Relief from chronic pelvic pain through surgical lesions of the conus medullaris dorsal root entry zone. Stereotact Funct Neurosurg. 1992;59(1-4):69-75. doi: 10.1159/000098920. PMID 1295050
- [Background] Howell B, Lad SP, Grill WM. Evaluation of intradural stimulation efficiency and selectivity in a computational model of spinal cord stimulation. PLoS One. 2014 Dec 23;9(12):e114938. doi: 10.1371/journal.pone.0114938. eCollection 2014. PMID 25536035
- [Background] Ranger MR, Irwin GJ, Bunbury KM, Peutrell JM. Changing body position alters the location of the spinal cord within the vertebral canal: a magnetic resonance imaging study. Br J Anaesth. 2008 Dec;101(6):804-9. doi: 10.1093/bja/aen295. Epub 2008 Oct 19. PMID 18936040
- [Background] Fettes PD, Leslie K, McNabb S, Smith PJ. Effect of spinal flexion on the conus medullaris: a case series using magnetic resonance imaging. Anaesthesia. 2006 Jun;61(6):521-3. doi: 10.1111/j.1365-2044.2006.04641.x. PMID 16704583
- [Background] Schultz DM, Webster L, Kosek P, Dar U, Tan Y, Sun M. Sensor-driven position-adaptive spinal cord stimulation for chronic pain. Pain Physician. 2012 Jan-Feb;15(1):1-12. PMID 22270733
- [Background] Parker JL, Karantonis DM, Single PS, Obradovic M, Cousins MJ. Compound action potentials recorded in the human spinal cord during neurostimulation for pain relief. Pain. 2012 Mar;153(3):593-601. doi: 10.1016/j.pain.2011.11.023. Epub 2011 Dec 19. PMID 22188868
- [Background] Mekhail NA, Levy RM, Deer TR, Kapural L, Li S, Amirdelfan K, Pope JE, Hunter CW, Rosen SM, Costandi SJ, Falowski SM, Burgher AH, Gilmore CA, Qureshi FA, Staats PS, Scowcroft J, McJunkin T, Carlson J, Kim CK, Yang MI, Stauss T, Petersen EA, Hagedorn JM, Rauck R, Kallewaard JW, Baranidharan G, Taylor RS, Poree L, Brounstein D, Duarte RV, Gmel GE, Gorman R, Gould I, Hanson E, Karantonis DM, Khurram A, Leitner A, Mugan D, Obradovic M, Ouyang Z, Parker J, Single P, Soliday N; EVOKE Study Group. ECAP-controlled closed-loop versus open-loop SCS for the treatment of chronic pain: 36-month results of the EVOKE blinded randomized clinical trial. Reg Anesth Pain Med. 2024 May 7;49(5):346-354. doi: 10.1136/rapm-2023-104751. PMID 37640452